CLINICAL TRIAL: NCT00004481
Title: Genetic Study of Sitosterolemia
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Medical University of South Carolina (Other)
Other Study IDs: NCRR-M01RR01070-0470; MUSC-HR-8022
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Lipid Metabolism, Inborn Errors; Sitosterolemia
Keywords: endocrine disorders; inborn errors of metabolism; rare disease; sitosterolemia
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Sitosterolemia; Endocrine System Diseases; Metabolism, Inborn Errors; Rare Diseases | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Natural History

INTERVENTIONS:
Procedure: genetic testing

SUMMARY:
OBJECTIVES:

I. Identify the genetic defect and fine map the gene that causes sitosterolemia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients, family members, and normal volunteers provide blood samples for genetic studies and may fill out a general health and medication history.

Linkage analysis and microsatellite screening is performed on genomic DNA, especially chromosome 2p21, between microsatellite markers D2S1788 and D2S1352.

Positive results may be reported to the patient and may influence future treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of sitosterolemia Presence of tendon and tuberous xanthomas Premature atherosclerotic disease No family history of premature coronary artery disease Normal or elevated plasma cholesterol levels

OR

* Family member of patient with sitosterolemia

OR

* Normal volunteer

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Shailesh B. Patel, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States